CLINICAL TRIAL: NCT04069923
Title: Use of Magnesium Oxide Biomaterial as a Bone Void Filler for Bone Voids or Defects Not Intrinsic to the Stability of Bony Structure
Brief Title: OsteoCrete in Filling Bone Voids in Participants With Bone Voids or Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-001785; NCI-2018-01668 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-001785 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2019-05-06; First posted 2019-08-28 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Health Status Unknown
MeSH Terms: interventions — OsteoCrete

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (OsteoCrete) (Experimental): Participants receive OsteoCrete intraoperatively to fill voids that occur in bones during surgery or to augment screw fixation.
  Interventions: Other: Magnesium-based Bone Void Filler

INTERVENTIONS:
Other: Magnesium-based Bone Void Filler — Given intraoperatively
  Other Names: Magnesium-based BVF; Osteocrete

SUMMARY:
This trial studies the side effects of OsteoCrete in filling bone voids in participants with bone voids or defects. OsteoCrete may eliminate the need for further surgery and the removal of healthy bone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of the device, which for the purpose of this study is defined as the compound injected into bone.

SECONDARY OBJECTIVES:

I. To determine the rate of absorption and bone ingrowth.

OUTLINE:

Participants receive OsteoCrete intraoperatively to fill voids that occur in bones during surgery or to augment screw fixation.

After completion of study treatment, participants are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of a diagnosis as evidenced by one or more clinical features consistent with one or more of the following criteria:

  * Bone void created during surgery.
  * Lucency noted on x-ray preoperatively.
* Written informed consent (and assent when applicable) obtained from subject or subject?s legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.
* Creatinine greater than 1.3.
* Presence of active bone infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Participants reaching one year post-op and completing all study visits | Up to 1 year

SECONDARY OUTCOMES:
Amount of reabsorption and bone ingrowth | Up to 1 year
  Will be measured in Hounsfield units by X-ray and compute tomography (CT).
Incidence of adverse events rates | Up to 1 year
  Will be coded by body system and MedDra classification term. Adverse events will be tabulated by treatment group and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study device.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Hornicek, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States